CLINICAL TRIAL: NCT05253378
Title: Development and Validation of a Comorbidity Index in Crohn's Disease
Acronym: NEMO-Index
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Dr Laurent PEYRIN-BIROULET, MD, PhD, Central Hospital, Nancy, France
Other Study IDs: 2021PI158
Record Dates: First submitted 2022-02-10; First posted 2022-02-23 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-05

CONDITIONS: Crohn Disease
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Crohn's disease (CD) is a chronic inflammatory bowel disease (IBD). Like other chronic diseases, patients with CD may be affected by other diseases called comorbidities. The prevalence of comorbidities in IBD patients ranges from 30 to 70 %. Unlike other chronic diseases, there is currently no CD-specific tool to assess the impact of comorbidities on patients' lives in order to take appropriate medical measures. Several clinical indexes have been developed for the study of comorbidities, including the Charlson index and the Groll index, which are widely used. The disadvantage of these indexes is that they are not adapted to patients with CD. The primary objective of this study is to develop and validate a clinical index to evaluate the impact of comorbidities on disability in patients with CD.

ELIGIBILITY:
Inclusion Criteria:

1. Patients between 18 and 59 years old
2. Established diagnosis of CD with a minimum disease duration of 3 months
3. Disease considered by the treating gastroenterologist to have been stable for at least 3 months

Exclusion Criteria:

1. Subject unable to comply with study procedures
2. Surgery for CD 3 months prior to inclusion visit

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: CD patients
Sampling Method: Non-Probability Sample
Enrollment: 458 (Actual)
Dates: Start 2022-04-04 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2025-03-31 (Actual)

PRIMARY OUTCOMES:
To develop and validate a clinical index to evaluate the impact of comorbidities on disability in patients with CD. | Through study completion, an average of 3 years
  Probability of having an IBD disability index ≥ 35 (i.e. moderate and severe disability).

CONTACTS AND LOCATIONS:
Locations (2):
- Laurent PEYRIN-BIROULET, Vandœuvre-lès-Nancy, France
- San Raffaele Hospital, Milan, Italy